CLINICAL TRIAL: NCT01752504
Title: Connect to Protect (C2P): Building a Community-Based Infrastructure for HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 095 - Version 3.0
Record Dates: First submitted 2011-07-08; First posted 2012-12-19 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-05

CONDITIONS: HIV Infection
Keywords: HIV prevention; HIV positive communities
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group (Experimental): Community members who become engaged in the coalitions and in the broader mobilization effort. A subset of community members..
  Interventions: Behavioral: Community Mobilization

INTERVENTIONS:
Behavioral: Community Mobilization — The proposed study seeks to continue C2P, a community mobilization intervention, which entails developing coalitions to plan for and bring about structural changes for purposes of reducing HIV incidence and prevalence among youth in targeted communities at five ATN sites. The C2P community mobilization model entails: determining a geographic area and population of focus for the coalitions to prioritize their planning and action; developing coalitions that have a shared vision and mission; developing a strategic plan focused on structural changes to reduce risks associated with HIV; documenting processes; providing feedback as technical assistance to the coalitions; hosting regular working group meetings; and on-going capacity building.

SUMMARY:
The proposed study seeks to continue the implementation of Connect to Protect® (C2P), a community mobilization intervention, which entails developing coalitions to plan for and bring about structural changes for purposes of reducing HIV incidence and prevalence among youth in targeted communities at five ATN sites.

DETAILED DESCRIPTION:
The C2P community mobilization model entails: determining a geographic area and population of focus for the coalitions to prioritize their planning and action; developing coalitions that have a shared vision and mission; developing a strategic plan focused on structural changes to reduce risks associated with HIV; documenting processes; providing feedback as technical assistance to the coalitions; hosting regular working group meetings; and on-going capacity building. The National Coordinating Center (NCC), operating under the direction of the Protocol Chair, provides guidance, training, technical assistance and feedback to coalitions.

The evaluation of C2P includes both process evaluation (i.e., documentation of coalition actions and achievements of structural changes; and outcome evaluation to qualitatively assess (via Key Informant (KI) interviews) if and how C2P efforts, including completed structural changes, have influenced the risk environment within each community. In addition, local health surveillance data and HIV testing data will be used to evaluate changes in HIV testing patterns and HIV/Sexually Transmitted Infection (STI) morbidity among youth.

ELIGIBILITY:
1. The intervention group = Community members who become engaged in the coalitions and in the broader mobilization effort; and
2. The evaluation group = Key Informants within each C2P community who either work or reside within the sectors or systems where structural changes have been accomplished and/or the coalition has focused their strategic planning efforts.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2011-11; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assess the extent to which C2P activities influence elements of the community that affect HIV-related risk prevention, testing, treatment and linkage to healthcare among youth aged 12-24 years and represent intermediate outcomes for this study. | End of year 5 (study completion)
  Assessment will include evaluation across three primary intermediate outcome areas:
  1. Achievement of Structural Change Objectives (SCOs) (programs, policies, practices) that target increased levels of HIV-related prevention, testing, and linkage to healthcare.
  2. Increased levels of community capacity and social capital to address HIV-related prevention, testing, and linkage to healthcare.
  3. Increased levels of sustainability across the HIV continuum of care (CoC) including prevention, testing, and linkage to healthcare activities initiated or influenced by C2P, including programs, policies, and new relationships

SECONDARY OUTCOMES:
Examine how attributes of the SCOs relate to intermediate outcomes in order to provide guidance and recommendations to policy makers. | End of year 5 (study completion)
  Attributes that will be analyzed include:
  1. Change strategy (e.g., information provisions, policy change, relationship formation, program creation).
  2. Sector(s) where change occurs.
  3. Distal and proximal causes targeted.
  4. Youth population affected by change (e.g., universal, selected, or indicated).
Assess the trends and associations with strategies used to achieve SCOs (e.g., creating linkages, honest brokering, strategic partnering, etc.) | End of year 5 (study completion)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ellen, MD, Study Chair — Johns Hopkins University Hospital
Locations (5):
- United States (5):
  - University of Colorado - The Children's Hospital of Denver, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Community Health, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: ATN Website — http://www.atnonline.org